CLINICAL TRIAL: NCT04182373
Title: A Phase 3, Randomized, Placebo-controlled, Double Blind Study of KW-3357 in Patients With Early Onset Severe Preeclampsia
Brief Title: KW-3357 Study in Patients With Early Onset Severe Preeclampsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Japan Blood Products Organization (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3357-101
Record Dates: First submitted 2019-10-10; First posted 2019-12-02 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Antithrombin
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KW-3357 (Experimental): 72 IU/kg
  Interventions: Drug: Antithrombin gamma
- placebo (Placebo Comparator)
  Interventions: Drug: physiological saline

INTERVENTIONS:
Drug: Antithrombin gamma — Intravenous infusion, once a day, 7 days
  Arms: KW-3357
Drug: physiological saline — Intravenous infusion, once a day, 7 days
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of intravenous KW-3357 in patients with early-onset severe preeclampsia by comparing the prolongation days of pregnancy with that of placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who gave written consent to participate in the clinical trial by their own free will.
2. Patients aged 18 years or older at the time of obtaining informed consent
3. Patients with early-onset PE* 24 weeks 0 days to 31 weeks 6 days of gestation at the time of enrollment

   *: Determine the definition of gestational age based on the ""Guidelines for Obstetrics and Gynecology, Obstetrics, 2020""
4. Patients diagnosed with severe PE*

   *: Follow the diagnostic criteria of the Japan Society for the Study of Hypertension in Pregnancy
5. Patients with AT activity of 100% or less in the preliminary examination

Exclusion Criteria:

1. Patients who are judged to require immediate delivery*

   *""Best Practice Guide 2015 for Care and Treatment of Hypertension in Pregnancy"" Requirements for Considering Pregnancy Termination Regardless of Pregnancy Weeks in Pregnancy-induced Hypertension Syndrome Cases will be consulted for judgment.
2. Patients with right hypochondralgia or epigastralgia
3. Patients with HELLP syndromes
4. Patients with pulmonary edema
5. Patients with severe pleural effusion, severe ascites, or serous retinal detachment
6. Patients with central nervous system disorders (eclampsia, stroke) or visual disorders (cortical blindness)
7. Patients with severe headache or urge eclampsia
8. Patients with abruptio placentae
9. Suspected patients with 8 or more obstetric DIC scores
10. Patients with a definitive diagnosis of congenital AT deficiency
11. Patients with diseases or symptoms other than the primary disease requiring immediate delivery
12. Patients on ongoing treatment with nonsteroidal anti-inflammatory drugs (NSAIDs, e.g., aspirin) or who require NSAIDs use during the course of the study.
13. Patients who have received the following drugs within 72 hours before administration of the investigational product, etc., or who require administration of the following drugs during the study period (from the start of administration of the investigational product, etc., until the date of termination of pregnancy); heparin, low-molecular-weight heparin (e.g., enoxaparin ordalteparin), fondaparinux, antiplatelet drugs (e.g., clopidogrel, prasugrel, aspirin), direct thrombin inhibitors (e.g., dabigatran), or anticoagulants (e.g., AT preparations).
14. Patients with a current or past history of serious drug allergy
15. Patients with a history or complication of drug dependence or alcoholism
16. Patients with hypersensitivity to AT preparations
17. Patients who are pregnant with a fetus with a chromosomal abnormality or a fetus suspected of having a serious malformation syndrome
18. Patients with multiple pregnancies
19. Patients with a history or complication of antiphospholipid antibody syndrome
20. Patients with diabetes complicated pregnancy or obvious diabetes mellitus
21. Patients with uncontrollable or significant complications, including the following

    * Clinically significant cardiovascular diseases, etc. (New York Heart Association cardiac function classifications Class III or higher)
    * Serious hepatic disease
    * Serious renal disease
    * Pneumonia, interstitial lung disease or other severe respiratory disease
    * Blood disorders such as idiopathic thrombocytopenic purpura
    * Psycho-central nervous system disorders that may affect informed consent
    * Endocrine disorders such as hyperthyroidism
    * Autoimmune diseases such as systemic lupus erythematosus
22. Patients with active malignancy or patients with a history of onset or treatment of malignancy within 5 years before pregnancy (excluding excised or surgically cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or ductal carcinoma of the breast, and excluding cervical intraepithelial neoplasia regardless of excised or surgically cured or not)
23. Patients with active infections (e.g., toxoplasma infection, genital chlamydia, genital herpes, cytomegalovirus infection)
24. Patients with a positive history for HIV antibody. Patients with a positive history for HBs antigen and HCV antibody and with active infection presenting with hepatitis symptoms.
25. Patients with any of the following laboratory abnormalities in preliminary examinations

    * Patients with AST or ALT 2 times the upper limit of the reference level of the trial site
    * Cr >=1.1 mg/dL
26. Patients who have participated in a clinical trial or equivalent study of a drug or medical device within 4 months before pregnancy (within 6 months for biologics) and have received the investigational drug or used an unapproved medical device
27. Other patients whom the principal investigator or the subinvestigator judges to be unfavorable for participation in the clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 181 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Days of maintaining pregnancy | Subjects will be observed until maternal and/or fetal indications for delivery necessitate cessation of expectant management or until approximately 34 0/7 weeks of gestation.

SECONDARY OUTCOMES:
Presence or absence of achievement of 32 weeks of gestation | 28 days before the end of study
Presence or absence of achievement of 34 weeks of gestation | 28 days before the end of study
Presence or absence of achievement of 28 weeks of gestation in subjects enrolled in the period of less than 28 weeks of gestation | 28 days before the end of study
Change in AT activity | From baseline to Day 8 at all time points and 3 days after termination of pregnancy
Change in PLT concentration | From baseline to Day 8 at all time points and 3 days after termination of pregnancy
Change on D-dimer concentration | From baseline to Day 8 at all time points
Change in FDP concentration | From baseline to Day 8 at all time points
Sitting systolic blood pressure and sitting diastolic blood pressure | From baseline to Day 8 at each time point, 3 days after termination of pregnancy, and 28 days after termination of pregnancy
Proteinuria/creatinine ratio | From baseline to Day 8 at each time point, 3 days after termination of pregnancy, and 28 days after termination of pregnancy
Amount of blood lost during delivery | 28 days before the end of study
Biophysical Profile Score | From baseline to Day 8 at each time point
  Minimum is 0, max is 10. Higher score means better condition.
Fetal growth rate | 28 days before the end of study
Apgar score | At 1 minute and 5 minutes after birth
  Minimum is 0, max is 10. Higher score means better condition.
Presence or absence of neonatal asphyxia | At 1 minute and 5 minutes after birth
Birth weight | 28 days before the end of study
Neonatal growth | 28 days before the end of study
  Fetal growth is classified into small for gestational age (SGA), appropriate for gestational age (AGA), and large for gestational age (LGA).
Head and chest circumferences at birth | 28 days before the end of study
Short-term prognosis of neonates (incidence of bronchopulmonary dysplasia, intraventricular hemorrhage, periventricular leukolame, retinopathy of prematurity, sepsis, necrotizing enteritis, death, etc) | 28 days after termination of pregnancy
The number of neonates who was hospitalized in the NICU | 28 days after termination of pregnancy
The number of days in the NICU | 28 days after termination of pregnancy
The number of neonates with respiratory management at the time of admission to the NICU | 28 days after termination of pregnancy
The number of days of respiratory management at the time of admission to the NICU | 28 days after termination of pregnancy

OTHER OUTCOMES:
Change in TNF-alpha at the time of examination | From baseline to Day 8
Change in interleukin (IL)-6 at the time of examination | From baseline to Day 8
Change in IL-10 at the time of examination | From baseline to Day 8
Change in hs-CRP at the time of examination | From baseline to Day 8
Change in sFlt-1 at the time of examination | From baseline to Day 8
Change in PlGF at the time of examination | From baseline to Day 8
Change in sFlt-1/PlGF at the time of examination | From baseline to Day 8
Pulsatility index of the umbilical artery and middle cerebral artery | At the time of examination from baseline to Day 8
Change in findings of the umbilical artery and middle cerebral artery | At the time of examination from baseline to Day 8
Distribution of reasons for termination of pregnancy | 28 days before the end of study
Prolongation days of pregnancy by reason of termination of pregnancy | 28 days before the end of study
Mode of delivery | 28 days before the end of study
Presence or absence of stillbirth | 28 days before the end of study. Neonates will be assessed after delivery.
Placental weight | 28 days before the end of study
Presence or absence of placental infarction | 28 days before the end of study
Umbilical arterial blood gas at termination of pregnancy | 28 days before the end of study
Presence or absence of HELLP syndromes and onset of symptoms | During the course of the clinical trial. Period from the day of commencement of administration of the investigational drug to Day 28 after the delivery

CONTACTS AND LOCATIONS:
Locations (63):
- Japan (63):
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Toyota Memorial Hospital, Toyota, Aichi-ken
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Tokyo Women's Medical University Yachiyo Medical Center, Yachiyo, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - National Hospital Organization Kokura Medical Center, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Our Lady of the Snow Social Medical Corporation St. Mary's Hospital, Kurume, Fukuoka
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Obihiro Kosei General Hospital, Obihiro, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Japanese Red Cross Society Himeji Hospital, Himeji, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Hizume, Iwate
  - National Hospital Organization Shikoku Medical Center for Children and Adults, Zentsujichó, Kagawa-ken
  - St. Marianna University School of Medicine, Kawasaki, Kanagawa
  - The Kitasato Institute Kitasato University Hospital, Sagamihara, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Sendai Red Cross Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto, Nagano
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - Nara Medical University Hospital, Kashihara, Nara
  - Okinawa prefectural Chubu Hospital, Uruma, Okinawa
  - Osaka Metropolitan University Hospital, Abeno-ku, Osaka
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Osaka Women's and Children's Hospital, Izumi, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Hamamatsu Medical Center, Hamamatsu, Shizuoka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - Dokkyo Medical University Hospital, Mibu, Tochigi
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Fuchū, Tokyo
  - Aiiku Hospital, Minato, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - National Center for Child Health and Development, Setagaya City, Tokyo
  - Japanese Red Cross Medical Center, Shibuya City, Tokyo
  - Showa University Hospital, Shinagawa, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Sumida City, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Aomori Prefectural Central Hospital, Aomori
  - Fukuoka University Hospital, Fukuoka
  - Kagoshima City Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Faculty of Medicine, University of Miyazaki Hospital, Miyazaki
  - Nagasaki University Hospital, Nagasaki
  - Nara Prefecture General Medical Center, Nara
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Oita Prefectural Hospital, Ōita
  - Toyama University Hospital, Toyama

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.

REFERENCES:
- [Background] Saito S, Takagi K, Moriya J, Kobayashi T, Kanayama N, Sameshima H, Morikawa M, Sago H, Adachi T, Ohkuchi A, Takeda S, Masuyama H, Seki H. A randomized phase 3 trial evaluating antithrombin gamma treatment in Japanese patients with early-onset severe preeclampsia (KOUNO-TORI study): Study protocol. Contemp Clin Trials. 2021 Aug;107:106490. doi: 10.1016/j.cct.2021.106490. Epub 2021 Jun 24. PMID 34174463